CLINICAL TRIAL: NCT04442841
Title: Hepatitis B Vaccination in Liver Transplant Reecipients Who Received a Liver From an Anti-core Positive Donor. H
Brief Title: HBV Vaccine in Anti-core Positive Donors After LT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: University of Padova (Other); Hospital Vall d'Hebron (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HBV Vaccine LT
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-06

CONDITIONS: Hepatitis B Reactivation
MeSH Terms: interventions — Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (vaccine) (Experimental): No further description
  Interventions: Biological: Hepatitis B vaccine

INTERVENTIONS:
Biological: Hepatitis B vaccine — It may be GSk or MSD vaccine

SUMMARY:
Anti-HBc positive liver donors frequently have occult HBV infection, and several studies in HBsAg-negative subjects have shown that there is often the detection in the liver of covalently closed circular DNA (cccDNA). In the setting of liver transplantation and immunosuppresion, grafts from antiHBc positive donors may cause de novo HBV infection (defined by the development of positive HBsAg and/or detectable serum or liver HBV DNA in previously HBsAg recipients).

Active immunization may be successful in up to 20% of patients who received an anti-HBc+ liver during transplantation after the first vaccination schedule, and up to 30% after a second vaccination course. Responders to vaccination could safely halt nucleos(t)ide analog prophylactic therapy with no risk of HBV reactivation during follow-up.

We also hypothesize that an impaired antigen-specific adaptive cell-mediated immunity at baseline explain the lack of response

Primary objective:

1. To investigate the efficacy of HBV vaccination in liver transplant recipients who received a liver from an anti-HBc positive donor.
2. To assess the safety of nucleos(t)ide treatment interruption in those patients achieving a response to HBV vaccination

DETAILED DESCRIPTION:
HYPOTHESIS The hypothesis of the study is that active immunization may be successful in up to 20% of patients who received an anti-HBc+ liver during transplantation after the first vaccination schedule, and up to 30% after a second vaccination course. Responders to vaccination could safely halt nucleos(t)ide analog prophylactic therapy with no risk of HBV reactivation during follow-up.

Thus, an impaired antigen-specific adaptive cell-mediated immunity at baseline may explain the lack of response.

OBJECTIVES

Primary objective:

1. To investigate the efficacy of HBV vaccination in liver transplant recipients who received a liver from an anti-HBc positive donor.
2. To assess the safety of nucleos(t)ide treatment interruption in those patients achieving a response to HBV vaccination

Secondary objectives:

1. To investigate which clinical and virological variables are associated with a protective response to HBV vaccination (including time from liver transplant, type of immunosuppressive therapy and vaccination prior liver transplantation)
2. To assess the role of HBV specific CD8 responses in developing a protective response to vaccination
3. To assess the relationship between intrahepatic cccDNA-HBV levels and the outcome after vaccination

   STUDY DESIGN This is a multi-center, open-label study in liver transplant recipients. Four transplant centers will include non-HBV liver transplant recipients who received a graft from an HBV anti-core positive donor. All patients should be under prophylactic nucleos(t)ide treatment (NA). Individuals will undergo HBV vaccination with double dosis vaccine (40 ug) and protective response will be evaluated at the end of a first course of vaccination. Response will be defined as anti-HBs levels > 100 IU/L. In patients who do not respond to a first course of vaccination, a second course will be administered.

   In patients achieving a protective immune response, prophylactic NA treatment will be interrupted and follow-up will be extended until 2 years after treatment interruption. Among those patients achieving vaccination response, a booster dose will be given if antiHBs levels fall below 100 IU/L during follow-up.

   Sample size calculation Sample size has been calculated in order to be able to identify variables that able to predict response/non response. The estimated number of anti-core positive recipients in all centers according to anti-core prevalence in general population is 160 patients (40 patients/center). According to previous reported data, around 20% would achieve a response to a first course of vaccination and an additional 30% would achieve response after a second course. With a confidance interval of 95% and accepting a precision level of 5% and an estimated loss rate of 15%, the calculated sample size would be 114 patients.

   Study flowchart All patients will receive 40 ug of HBV vaccine, at 0, 1 and 3 months time points.

   In patients not achieving protective anti-HBs titers (≥ 100 IU/L) 1 month after the last HBV vaccine dose, the same vaccine schedule will be repeated (40 ug of vaccine 0, 1 and 3 months).

   Patients not achieving protective anti-HBs titers (≥ 100 IU/L) 1 month after last HBV vaccine dose will be considered non-responders and will continue on NA therapy.

   In patients achieving protective anti-HBs titers, prophylaxis with nucleoside analogues will be interrupted and patients will be followed for a minimum period of 24 months. Blood tests will be performed every 6 months including liver tests, markers of HBV reactivation and anti-HBs. If anti-HBs levels fall below <100 IU/L at any time point of follow-up, a single boost (40 ug) will be repeated.

   In case of HBV reactivation (HBsAg or HBV-DNA positive) during follow-up, oral NA therapy will be restarted with high barrier to resistance drugs such as entecavir or tenofovir.

   Study procedures All patients Screening visit
   * Medical history and physical examination.
   * Review inclusion and exclusion criteria.
   * Obtain written informed consent.
   * Complete blood tets

     * Hematology, chemistry and coagulation tests.
     * Serologies: HBsAg, IgG HBV anti-core (HBc), anti-HBs, HIV antibody, IgG HCV
     * HBV-DNA, HCV-RNA (only if anti-HCV positive)
     * Liver biopsy (if the patient signs an additional inform consent)
   * Extraction of 40 ml of blood to process PBMC (Hospital Clínic Barcelona and Padova University Hospital)
   * Liver Biopsy (Hospital Clínic Barcelona) in order to exclude the presence of liver fibrosis (or other lesions) and to obtain frozen tissue and evaluate the presence of cccDNA and its correlation with study outcomes.

   Baseline (day 1):

   The following procedures will be completed prior to treatment administration:
   * Perform a complete physical examination.
   * Extraction of 40 ml of blood to process PBMC Thereafter, the first dose of vaccine (GSK 40 ug) will be administered Week 4: 2nd dose of vaccine Week 12: 3rd dose of vaccine

   Week 16:
   * Medical history and physical examination.
   * Complete blood tets

     * Hematology, chemistry and coagulation tests.
     * Serologies: HBsAg, anti-HBc, anti-HBs,
     * HBV-DNA
   * Extraction of 40 ml of blood to process PBMC (Hospital Clínic Barcelona and Padova University Hospital) a) Responders If anti-HBs ≥ 100 IU/L Interruption of nucleoside analogue* (in patients who qualify for NA interruption, a specific follow-up will continue, as described below) b) Non-responders If anti-HBs < 100 IU/L First dose of second course of vaccination Week 20: 2nd dose of vaccine Week 32: 3rd dose of vaccine

   Week 38:
   * Medical history and physical examination.
   * Complete blood tets o Hematology, chemistry and coagulation tests.

     o Serologies: HBsAg, anti-HBc, anti-HBs,

     o HBV-DNA
   * Extraction of 40 ml of blood to process PBMC (Hospital Clínic Barcelona and Padova University Hospital)

     1. Responders If anti-HBs ≥ 100 IU/L Interruption of nucleoside analogue (in patients who qualify for NA interruption, a specific follow-up will continue, as described below)
     2. Non-responders If anti-HBs < 100 IU/L will continue NA therapy

        * Responders to vaccination and NA withdrawal: follow-up every 2 months during the first 6 months and every 6 months until 2 years of follow-up

   At each visit:

   Medical history and physical examination.

   Complete blood tets:

   o Hematology, chemistry and coagulation tests.
   * Serologies: HBsAg, Anti-HBs
   * HBV-DNA If anti-HBs < 100 IU/L : a vaccine booster (40 ug) will be administered If HBsAg+ or HBV-DNA+ confirmed in two occasions 2 weeks apart: NA therapy with entecavir or tenofovir will be introduced.

   Statistical analysis Statistical analysis will be performed using SPSS, version 22 (SPSS, Chicago, IL). Categorical data will be analyzed using the chi-square test; continuous data will be analyzed using the Student T test. The survival rates were calculated using the Kaplan-Meier method with log- rank test for significance. A P value of<0.05 will be considered

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years- old.
* HBsAg-negative pre-transplantation
* Liver transplant recipients; more than 2 years from the date of LT
* Transplantation of a graft from an HBV anti-core positive donor
* Patients should be under nucleoside analogue therapy with Lamivudine, Tenofovir or Entecavir
* Stable immunosuppressive therapy during the last 6 months
* Baseline anti-HBs levels <100 IU/L (HBV vaccination while on the waiting list is allowed and will be recorded)
* Willingness to participate in the study and written inform consent

Exclusion Criteria:

* • HBsAg positive at any time post-transplantation

  * HBV-DNA positive at any time post-transplantation
  * Any HBIG dose during the last 12 months
  * HBV vaccination after liver transplantation
  * Spontaneous or vaccine-induced post-transplant anti-HBs titers ≥ 100 UI/L
  * Any rejection episode during the last 12 months
  * Positive HCV-RNA at time of vaccination
  * HCV therapy with direct acting antivirals within the previous 12 months
  * HIV coinfection
  * Advanced fibrosis after LT (liver stiffness measurement ≥ 9.5 kPa)
  * Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Response to HBV vaccine | 1 month after last HBV vaccine dose
  > 100 IU/mlL anti-HBs
Incidence of Emergent Adverse Events in case of nucleos(t)ide analogue (NUC) treatment interruption | 6 months after NUC interruption
  No reactivation of HBV (negative HBV-DNA) 6-12 months after NUC interruption

CONTACTS AND LOCATIONS:
Locations (1):
- Liver Unit, Hospital Clinic, Barcelona, Spain